CLINICAL TRIAL: NCT00852722
Title: A Randomized, Controlled Study of Diet and Multiple Sclerosis
Brief Title: Low Fat Diet and Multiple Sclerosis
Acronym: MS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Vijayshree Yadav, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OHSU IRB00004555
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Diet
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Low fat study diet (Experimental): The low fat study diet arm will receive low fat diet training and followed for 12 months on the diet.
  Interventions: Other: Low fat study diet
- 2. Regular diet group (No Intervention): The regular diet arm will be a wait-listed group that will receive no training in diet and will be advised to continue their regular (usual) diet as was prior to entry into the study, for the duration of the study. They will have a similar clinic follow up schedule as the treatment group. The regular diet group will be given identical instructions to exercise regularly similar to the treatment group.

INTERVENTIONS:
Other: Low fat study diet — The low fat study diet is a very low-saturated-fat, plant food based diet. It will be approximately 10% fat, 14% protein and 76% carbohydrate.The diet is is starched based and also contains fresh or frozen fruits and vegetables and there is no animal meat used, including no use of fish. This diet is very low in saturated fats and enriched in unsaturated fats. Subjects do not take dietary supplements.
  Arms: 1. Low fat study diet

SUMMARY:
The purpose of this study is to evaluate if following a specific low fat diet will improve the brain damage as seen by Magnetic Resonance Imaging (MRI) and to decrease the progression of multiple sclerosis (MS) as evidenced by clinical evaluation and symptoms.

DETAILED DESCRIPTION:
This research project has significance for its potential to develop a new therapeutic approach to MS. Current treatments in MS include disease modifying therapies such as human recombinant interferon beta, glatiramer acetate and natalizumab. However, these are only partially effective, cannot be taken orally, have side-effects and are very expensive. Developing treatment that can be combined with current disease modifying agent remains an important goal for improving the care of people with MS.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of the relapsing-remitting form of MS
* Age 18-70, inclusive
* MS duration of less than 15 years
* May or may not be on disease-modifying therapies for MS, but if on, must be on for more than 6 months of continuous therapy
* Should not have diabetes
* Able and willing to follow exercise instructions
* Able and willing to travel to California for 10-day training program (cost covered by study)
* Able and willing to travel to Portland, OR for 6 study visits over the 12 month study period (cost covered by study)

Exclusion Criteria:

* No clinically significant MS exacerbation within 30 days of screening visit
* No systemically administered corticosteroids within 30 days of study entry
* Patient not pregnant or breastfeeding
* Not taking fish oil/flax seed for at least 2 months prior to first visit
* No other significant health programs (e.g. active coronary heart disease, liver disease, pulmonary disease) that might increase risk of patient experiencing adverse events

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of new MS T2 lesion formation on brain MRI in those randomized to the low fat study diet with that of subjects randomized to follow their regular diet. | Baseline. Month 12.

SECONDARY OUTCOMES:
To assess effects of the low fat study diet on clinical activity of MS as by relapse rate and disability progression and on fatigue, depression and quality of life. | Baseline. Month 3. Month 6. Month 9. Month 12.
To study the effects of the Low Fat Study Diet on serum markers of inflammation | Baseline. Month 6. Month 12.
To assess safety and tolerability of the low fat study diet upon 12 months of administration | Baseline. Month 3. Month 6. Month 9. Month 12.

CONTACTS AND LOCATIONS:
Overall Officials: Vijayshree Yadav, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- See also: MS Center of OHSU website — http://www.ohsu.edu/ms